CLINICAL TRIAL: NCT02468609
Title: Diagnostic Value of Ultralow-dose Computed Tomography for the Detection of Pulmonary Nodules and Lung Parenchym Alterations Compared to Standard-dose CT
Acronym: RADFL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Michael Messerli, MD, Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: EKSG 15/007
Record Dates: First submitted 2015-01-30; First posted 2015-06-11 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Pulmonary Nodules; Pulmonary Emphysema
MeSH Terms: conditions — Multiple Pulmonary Nodules; Pulmonary Emphysema

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultralow-Dose-CT (Other): Additional Ultralow-Dose-CT of the chest
  Interventions: Radiation: Ultralow-Dose-CT

INTERVENTIONS:
Radiation: Ultralow-Dose-CT — Patients undergoing thoracic normal dose-CT with undergo an additional Ultralow-Dose-CT

SUMMARY:
To investigate the diagnostic value of ultralow-dose computed tomography in the detection of pulmonary nodules and lung parenchym alterations (e.g. emphysema) compared to standard-dose-CT.

ELIGIBILITY:
Inclusion Criteria:

* planned normal dose-CT by clinical indication at our institution
* obtained informed consent

Exclusion Criteria:

* planned lowdose-CT by clinical indication at institution
* no informed consent obtained
* age < 18 years
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of pulmonary Nodules detected in the Ultralow-Dose thoracic CT | Participants CT-scan will be read out on an average date of 6 weeks after the scan
  Difference in nodule detectability in Ultralow-Dose-CT compared to Standard-Dose-CT measured using McNemar test

SECONDARY OUTCOMES:
Patients BMI (Body mass index) | Measures assessed at time of read-out on an average date of 6 weeks after the scan
Patients Nodule size (mm) | Measures assessed at time of read-out on an average date of 6 weeks after the scan

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Radiologie und Nuklearmedizin, Sankt Gallen, Switzerland